CLINICAL TRIAL: NCT05666726
Title: State-Dependent Interoception, Value-Based Decision Making, and Introspection
Brief Title: State-dependent Interoception, Value-based Decision-making, and Introspection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10000978; 000978-M
Record Dates: First submitted 2022-12-27; First posted 2022-12-28 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01-22

CONDITIONS: Stress; Pain; Emotions; Craving; Frustration
Keywords: Decision-Making; Interoception; Metacognition; Stress; Pain; Negative Emotion
MeSH Terms: conditions — Pain | interventions — Projective Techniques

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1 (Experimental): within-subjects experimental study, where each subject will receive a neutral state and a negative state induction intervention in a cross-over design (counterbalanced order across participants).
  Interventions: Behavioral: Negative valence emotion
- 2 (Experimental): within-subjects experimental study, where each subject will receive a neutral state and a negative state induction intervention in a cross-over design (counterbalanced order across participants).
  Interventions: Behavioral: Frustration
- 3 (Experimental): within-subjects experimental study, where each subject will receive a neutral state and a negative state induction intervention in a cross-over design (counterbalanced order across participants).
  Interventions: Other: Pain
- 4 (Experimental): within-subjects experimental study, where each subject will receive a neutral state and a negative state induction intervention in a cross-over design (counterbalanced order across participants).
  Interventions: Other: Stress
- 5 (Experimental): within-subjects experimental study, where each subject will receive a neutral state and a negative state induction intervention in a cross-over design (counterbalanced order across participants).
  Interventions: Behavioral: Craving

INTERVENTIONS:
Other: Pain — Thermal pain
  Arms: 3
Other: Stress — Stress state induction
  Arms: 4
Behavioral: Craving — Snack craving induction
  Arms: 5
Behavioral: Frustration — Real effort task
  Arms: 2
Behavioral: Negative valence emotion — Passive video watching with emotional valence
  Arms: 1

SUMMARY:
Background:

Negative emotional states can affect a person s behavior as they make decisions. For example, hunger may make people more impatient; they may then make riskier choices. Other negative emotional states that can change behavior include stress, pain, and sadness. By learning more about how emotions affect thinking and behavior in healthy people, researchers hope to better understand how to identify and treat people with mental disorders.

Objective:

To learn how negative emotions affect the brain and decision-making behavior.

Eligibility:

Healthy people aged 18 to 55 years.

Design:

Participants will have 3 clinic visits in 3 weeks.

Participants will fill out questionnaires. They will be asked about their personal history, their personality, and state of mind.

For 2 visits, participants will be assigned to different groups. Each group will experience 1 type of emotional stressor:

Some participants will watch a video.

Some will have to do arithmetic problems.

Some will have heat applied to an arm or leg.

Some will experience cold by immersing their hand in ice water.

For a snack craving test, some will be tempted by food after a 4-hour fast.

During these tests, participants will have sensors attached to their bodies. They will be videotaped. Saliva samples will be collected.

After the stressors, participants will do tasks on a computer. They will need to make choices.

Some participants will perform these decision-making tasks while lying in a brain scanner for functional magnetic resonance imaging. The brain scan involves lying on a table that slides into a cylinder that takes images of the brain.

...

DETAILED DESCRIPTION:
Study Description:

This study involves a series of experiments consisting of within-subject experimental manipulations of state. In separate sub-studies, we will induce 5 types of negative valence states (negative emotion, loss, pain, stress, and craving) compared to a neutral state to test the hypothesis that negative valence states impact value-based decision-making and the neural mechanisms involved in decision-making.

Objectives:

Primary Objective: Determine the effect of induced negative valence states on value-based decision-making and examine how brain value representation during decision-making is affected by negative valence states.

Secondary Objectives: 1) Determine the role of interoception and metacognition as moderators of the effect of negative valence states on value-based decision-making. 2) Characterize state-specific effects on value-based decision-making. 3) Establish whether states can affect stable features of interoception and metacognition. 4) Build a classification model for state-specific detection using multimodal feature data. 5) Compare interoception across modalities (cardiac, respiratory, pain). 6) Characterize state-specific neuroendocrine profiles for gonadal, stress, and appetitive hormones. 7) Explore how psychological stress and negative affect alter self-reported enjoyment in value-based actions.

Endpoints:

Primary Endpoints: Choice behavior and brain activations in decision-making tasks: 1) willingness-to-pay, 2) risk aversion, 3) ambiguity

aversion, and 4) delay discounting. For fMRI: 1) VMPFC BOLD, 2) VS BOLD, and 3) AI BOLD signal.

Secondary Endpoints: Behavior and neural activations in an interoceptive task and confidence reports: 1) interoceptive accuracy, 2) confidence bias, and 3) confidence sensitivity. Behavior and neural activations in an enjoyable goal-progress task and pleasure reports: 1) local goal progress, 2) pleasure experience. For fMRI: 1) OFC BOLD, 2) vmPFC BOLD, 3) ACC BOLD, 4) VS BOLD, 5) network

connectivity.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subject selections will be equitable among those individuals who meet the inclusion criteria. Every effort will be made to balance sex and race. In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Ability of subject to understand and the willingness to sign a written informed consent document.
* All sexes; Age 18 to 55.
* Able to read and write in English to guarantee understanding of all written and spoken instructions, which are in English.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

For all experiments:

* Unable to comply with study procedures or follow-up visits
* Has any serious or unstable medical condition or history that in a clinician s assessment implies a cardiovascular, neurological, or physical risk from the study procedures performed to induce negative valence states. This may include chronic systemic disorders that could worsen due to stress (e.g. uncontrolled hypertension, coronary artery disease for example a history of myocardial infarction or stable or unstable angina, or diabetes)
* Has any current psychiatric diagnosis (based on SCID or the MINI Mini International Neuropsychiatric Interview) or no diagnosis but scores >=29 on Beck Depression Inventory II or >=26 on Beck Anxiety Inventory
* Meets criteria for diagnosis of any substance-related or addictive disorder, or endorses any kind of problematic gambling behavior or problematic media-based addictive behavior (such as videogames, social-networking, online shopping, etc.)
* Regular use of psychoactive medications or psychoactive substances
* Regular use of corticosteroids
* Is pregnant

For stress and pain induction:

* Has a major medical condition or medical history that in a clinician s assessment could affect temperature sensitivity, pain thresholds, or ability to comply with study procedures. This may include cardiovascular, autonomic, neurological, psychiatric, or chronic systemic disorders (including but not limited to stroke, blindness, deafness, history of brain damage, neurodegenerative, neurotoxic or demyelinating disorder, or diabetes)
* Has a medical condition that in a clinician s assessment might affect somatosensation (e.g., Raynaud s disease, peripheral neuropathy, or circulatory disorder)

For pain induction:

* Has a current chronic pain condition or has had chronic pain in the past (painful condition lasting more than six months)
* Has a dermatological condition such as scars or burns, or has had a tattoo in the testing region within the previous 4 weeks that might influence cutaneous sensibility
* Regular and recent use of prescription or over-the-counter medication that has a significant effect on pain or heat perception. These include medications such as centralacting agents such as opiates (morphine, tramadol), antidepressants (amitriptyline, duloxetine, milnacipran), anticonvulsants (gabapentin, pregabalin), anxiolytics (barbiturates, benzodiazepines), hypnotics (zolpidem, sodium oxybate), antipsychotics (valproate, lithium, olanzapine), antimigraine agents (sumatriptan, ergotamine), and muscle relaxants (cyclobenzaprine, carisoprodol). Use of analgesic medications, such as non-steroidal anti-inflammatories, salicylates, and acetaminophen, taken on an as needed basis is acceptable as long as the last dose taken was within 5 half-lives of testing.

For craving induction:

* Has a condition that in a clinician s assessment could preclude the ability to hold 4-6 hours of fasting or that is associated with a risk of hypoglycemia (such as diabetes, kidney disease, insulinoma, adrenal or pituitary tumors or disorders, or anorexia nervosa)
* Is currently engaged in any kind of diet medically- or self-prescribed or endorses a very strong desire to start a diet that involves eliminating or decreasing carbohydrate consumption
* Has a history of food allergies such as tree-nut or peanut allergy.

For fMRI experiments:

* Individuals with conditions that could pose a risk relating to the safety of the fMRI procedure but do not meet specific exclusion criteria for all experiments or for specific inductions will be excluded from the MRI portion of the protocol but may participate in the non-MRI sessions. Such conditions include:
* Those with ferromagnetic metal in the cranial cavity or eye (e.g. aneurysm clip, implanted neural stimulator, cochlear implant, ocular foreign body)
* Those with an abnormality on a structural MRI
* Those with an implanted cardiac pacemaker or auto-defibrillator
* Those with an insulin pump
* Those with an irremovable body piercing
* Pregnancy (based on urine test completed within 24 hours prior to scan)
* Left-handed (only for fMRI experiments involving thermal pain stimulation)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 900 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Value-based decision-making metrics | Right after intervention
  Value-based metrics such as delay discounting, which is a measure of an individual's preference for small immediate rewards over larger later rewards.
BOLD signal in decision-making areas ROI | Right after intervention
  BOLD signal related to decision making tasks

SECONDARY OUTCOMES:
Confidence | Right after intervention
  Level of confidence on the accuracy or optimality of their behavior.
Interoceptive accuracy | Right after intervention
  Interoceptive accuracy is a measure of an individual's ability to report on bodily sensations with precision.

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Lopez Guzman, M.D., Principal Investigator — National Institute of Mental Health (NIMH)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. @@@@@@@@@@@@All individual participant data that underlie results in a publication will be made publicly available. No Personal Identifiable Information will be shared, all data submitted to repositories will be deidentified.
Supporting Information: SAP
Time Frame: Data from this study may be requested from other researchers 1 year after the completion of the primary endpoint by contacting the NIMH Data Archive (NDA) for all behavioral data and OpenNeuro (www.openneuro.org) for all fMRI data. It will remain in said repositories indefinitely.
Access Criteria: All individual participant data that underlie results in a publication will be made public through the IMH Data Archive (NDA) and OpenNeuro (www.openneuro.org) repositories. Access criteria is defined by these repositories and will not be limited by analysis type.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000978-M.html